CLINICAL TRIAL: NCT02243488
Title: Does Menstrual Hygiene Matter? Randomised Control Step-Wedge Trial Investigating the Impact of a Menstrual Hygiene Program (Reusable Sanitary Pad and Menstrual Health Education) on Rural Ugandan Girls' School Absenteeism
Brief Title: Does Menstrual Hygiene Matter? Investigating the Impact of a Menstrual Hygiene Program on Ugandan Girls' School Absenteeism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irise International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0677/KW; SAS-2014-010\7 (Other Grant/Funding Number: The Leverhulme Trust)
Record Dates: First submitted 2014-09-05; First posted 2014-09-18 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Menstrual Hygiene Management
Keywords: Menstruation; MHM; Menstrual Hygiene Management; Girls Education; Absenteeism; Access to Education; Menstrual Health Education; Reusable Sanitary Product

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12 month menstrual hygiene programme (Experimental): This is the first group to receive the intervention. They will receive the intervention after baseline and be followed up for the following 12 months.
  Interventions: Device: Irise Easy Pad & Menstrual Health Education
- 6 month menstrual hygiene programme (Experimental): This is the second group to receive the intervention. They will act as a control group for the first 6 months then receive intervention at 6 months.
  Interventions: Device: Irise Easy Pad & Menstrual Health Education

INTERVENTIONS:
Device: Irise Easy Pad & Menstrual Health Education — Reusable manufactured sanitary pad produced by Irise Uganda Limited and education sessions provided by qualified menstrual health educators

SUMMARY:
This study builds on the pilot work of the Irise research group to investigate the impact of menstrual hygiene interventions on East African girls' school attendance, activities of daily living and self-esteem. The trial will be carried out in 40 schools to either intervention or control arms. Schools will receive a menstrual hygiene program, including the distribution of reusable sanitary pads and menstrual health education. The impact of the programme on girls' school attendance will be monitored using the validated Irise questionnaire and school registers. The impact of the programme on activities of daily living during menstruation and self-esteem during menstruation will also be measured using the Irise Questionnaire and explored using focus groups.

DETAILED DESCRIPTION:
Research Aims and Objectives

Aims

- To assess the impact of a Menstrual Hygiene Management (MHM) Programme, based around the distribution of reusable pads and delivery of health education in schools, on East African schoolgirls.

Objectives

* To explore initial (baseline) MHM practices and knowledge
* To assess school absenteeism during the study period
* To assess the impact of menstruation on activities of daily living at baseline and at 6 and 12 months into the study
* To assess girls' self-esteem during menstruation at baseline and at 6 and 12 months into the study

Background

Irise International

Irise International is a small charitable organisation and research group founded in 2011 in response to Kenyan school girls' accounts of their difficulties attending school during menstruation. School enrolment in East Africa is the highest it has ever been. In Uganda primary school enrolment is 94% with almost equal numbers of girls and boys enrolled in the first grade. However primary school completion rates are only 25% for girls, compared to 56% for boys. This data highlights a need for interventions to help keep girls in school so they can make the most of the opportunities they are being offered. It is in this context that menstrual hygiene and sanitation interventions may become an important means of promoting girls' education and empowerment.

Pilot work

Irise undertook a pilot study in Kisumu Kenya. Groups of 30 girls from 10 schools were randomly allocated to control or intervention groups. The intervention group received training on how to make a reusable pad and enough equipment to make three. Data was collected at baseline and at one month using a questionnaire. The mean number of days girls reported missing specifically due to menstruation was 1.66 with responses ranged from 0-11. Overall 5 in 10 girls reported missing some school because of menstruation compared to just 1 in 10 in the UK.

After one month follow-up, absenteeism was reduced, on average, by 1.5 days in the schools that received the intervention. A covariate adjusted t-test of group mean number of days missed, control group vs intervention group, showed a result that was close to the 95% significance level (2.01 mean days (±2.14) vs 1.32 mean days (±1.89); P=0.077; 95% CI -3.17: 0.21).

For all schools in the intervention group the mean number of days of school missed decreased or stayed constant; schools in the control group either stayed constant or increased.

More research is needed to investigate the long term effect of menstrual hygiene programmes on school girls' attendance, activities of daily living and self-esteem. This study will therefore build on the investigators previous pilot work and is part of an on-going process to research this neglected issue.

Preliminary work

A preliminary round of data collection took place in June and July 2013 in 30 schools through the delivery of a questionnaire. A more detailed investigation using interviews was carried out in a select number of schools in order to understand local menstrual hygiene practices in more depth and collect context specific information relevant to the delivery of a menstrual hygiene program. It also enabled us to introduce the concept of research and how it should be conducted to the investigators local partner and helped to identify logistical issues which the investigators can take steps to avoid in the main study.

Research methods

Design

A step wedge design was chosen to provide a control group for 6 months but allow all girls enrolled in the study to receive the intervention at 12 months. The investigators will also be able to see if the effect of the intervention in the intervention group is replicated in the control when they receive the intervention at six months. Class 6 in each school will be enrolled in the study and will receive pads and menstrual health education. Schools will be selected a predefined distance apart in order to avoid contamination. If schools do fall less than the predefined distance apart they will be classed as a cluster and be analysed together. At baseline half the schools will be randomly allocated to receive the intervention and while the other half will act as a control group. After six months the remaining schools will also be given the intervention and all schools will be followed up for the remainder of the study period.

Recruitment of schools

Forty schools in Western Uganda will be recruited through local Irise partner, LuYoDeFo and through contacts at Kampala International University and the Department of Health. These Irise partners and contacts will provide a list of schools in the areas selected to take part in the research. These schools will then be visited by an Irise researcher and be given information about the study. They will have the opportunity to opt in or out at this point. Written informed consent will be obtained from the head teachers of the schools and from the girls themselves.

Planned Intervention

During the first 6 months 20 schools will receive menstrual health education and free promotional reusable pads from a local social enterprise set-up as part of Irise's project work in Uganda. During the second 6 months the remaining 20 schools will receive menstrual health education and free promotional pads from the local social enterprise.

ELIGIBILITY:
Inclusion Criteria:

* Girls from schools who have not previously been recipients of a menstrual hygiene programme between the ages of 14-18 who have started menstruating.

Exclusion Criteria:

* Girls who have not started their periods will be excluded.

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The number of days of school missed per month | Baseline
  The number of days of school missed during a month for the female members of the class in the participating school. This will be measured through self-reported questionnaires and the results will be triangulated through the use of school registers.
The number of days of school missed per month | Baseline to 6 months
  The number of days of school missed during a month for the female members of the class in the participating school. This will be measured through self-reported questionnaires and the results will be triangulated through the use of school registers.
The number of days of school missed per month | 6 months to 12 months
  The number of days of school missed during a month for the female members of the class in the participating school. This will be measured through self-reported questionnaires and the results will be triangulated through the use of school registers.

SECONDARY OUTCOMES:
Impact of menstruation on activities of daily living | Baseline
  This will be measured through self-reported questionnaires. The questions are part of the validated questionnaire developed by Irise International on menstrual hygiene. The frequency that menstrual hygiene interferes with participants ADLs can be categorized. Proportions can then be displayed to give an idea of impact.
Impact of menstruation on activities of daily living | 6 months
  This will be measured through self-reported questionnaires. The questions are part of the validated questionnaire developed by Irise International on menstrual hygiene. The frequency that menstrual hygiene interferes with participants ADLs can be categorized. Proportions can then be displayed to give an idea of impact.
Impact of menstruation on activities of daily living | 12 months
  This will be measured through self-reported questionnaires. The questions are part of the validated questionnaire developed by Irise International on menstrual hygiene. The frequency that menstrual hygiene interferes with participants ADLs can be categorized. Proportions can then be displayed to give an idea of impact.
Self-esteem during menstruation | Baseline
  The impact of menstruation on participants self-esteem will be investigated through qualitative techniques of focus groups and interviews.
Self-esteem during menstruation | 6 months
  The impact of menstruation on participants self-esteem will be investigated through qualitative techniques of focus groups and interviews.
Self-esteem during menstruation | 12 months
  The impact of menstruation on participants self-esteem will be investigated through qualitative techniques of focus groups and interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Wilson-Smith, BA, MBChB, Principal Investigator — Irise International
Locations (1):
- Kampala International University, Kasese, Kasese, Uganda

REFERENCES:
- [Background] Emily Wilson, Josephine Reeve & Alice Pitt Education. Period. Developing an acceptable and replicable menstrual hygiene intervention Development in Practice 24(1): 63-80, 2014
- See also: Related Info — http://www.irise.org.uk